CLINICAL TRIAL: NCT06099977
Title: The Effect of Preoperative Binaural Sound on Remimazolam Dose Required for Induction of General Anesthesia: a Randomized, Placebo-controlled Trial
Brief Title: Binaural Sound for Remimazolam Induction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Clinical Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 3-2023-0305
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: General Anesthesia; Prostate Cancer; Uterine Myoma
MeSH Terms: conditions — Prostatic Neoplasms; Myofibroma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Binaural) (Experimental): Binaural sound using headphone will be applied.
  Interventions: Procedure: Binaural sound
- II (Placebo) (Placebo Comparator): Only headphone without sound will be applied.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Binaural sound — Binaural sound: Binaural sound will be applied.
  Arms: I (Binaural)
Procedure: Placebo — Only headphone without sound will be applied.
  Arms: II (Placebo)

SUMMARY:
It is important to decrease the time-to-loss of consciousness and anesthetics dose of remimazolam for general anesthesia induction. We will evaluate the effect of binaural sound for general anestheia induction using remimazolam infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for generla anesthesia
2. Patients aged 20-60
3. Patients with American Society of Anesthesiologist physical status classification 1-2
4. Patients with ideal body weight 50-80 kg

Exclusion Criteria:

1. Patients with hearing disability
2. Patients using opioids or sedatives in 1 week
3. Patients who are dependent for alcoholics or drugs
4. Patients with hypersensitivities to remimazolam
5. Patients with arrhythmia, cardiovascular disease, heart failure, or hypovolemia
6. Patients with liver failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Remimazolam dose for no response to voice | At anesthesia day 0
  Remimazolam dose for no response to voice will be measured at anesthesia day 0.

SECONDARY OUTCOMES:
Remimazolam dose for no eye lash reflex | At anesthesia day 0
  Remimazolam dose for no eye lash reflex will be measured at anesthesia day 0.
Remimazolam dose for patient state index 50 | At anesthesia day 0
  Remimazolam dose for patient state index 50 will be measured at anesthesia day 0.
Anxiety level | At anesthesia day 0
  Anxiety level will be evaluated using viosual analogue scale at anesthesia day 0 (at arrival of preanesthetic room and operating room).
Patient state index electroencephalography | At anesthesia day 0
  Patient state index electroencephalography will be evaluated at anesthesia day 0

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeveranceHospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided